CLINICAL TRIAL: NCT06122714
Title: A Phase I Randomised, Single-blind, Placebo-controlled, and Sequential Group Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD4144 Following Single and Multiple Ascending Doses Via Oral Administration to Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD4144 Following Single and Multiple Ascending Doses Via Oral Administration to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D9440C00001
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Healthy Participants
Keywords: Single ascending dose (SAD); Multiple ascending dose (MAD)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Part A1 (healthy participants) Cohort 1 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A1 (healthy participants) Cohort 2 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A1 (healthy participants) Cohort 3 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A1 (healthy participants) Cohort 4 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A1 (healthy participants) Cohort 5 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A1 (healthy participants) Cohort 6 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A1 (healthy participants) placebo (Placebo Comparator): Participants will receive matching Placebo.
  Interventions: Drug: Placebo Part A
- Part A2 (healthy Japanese participants) Cohort 1 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A2 (healthy Japanese participants) Cohort 2 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A2 (healthy Japanese participants) placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo Part A
- Part A3 (healthy Chinese participants) Cohort 1 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part A
- Part A3 (healthy Chinese participants) placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo Part A
- Part B1 (healthy participants) Cohort 1 (Experimental): Participants will receive one multiple ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part B
- Part B1 (healthy participants) Cohort 2 (Experimental): Participants will receive one multiple ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part B
- Part B1 (healthy participants) Cohort 3 (Experimental): Participants will receive one multiple ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part B
- Part B1 (healthy participants) placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo Part B
- Part B2 (healthy Japanese participants) Cohort 1 (Experimental): Participants will receive one multiple ascending dose of AZD4144.
  Interventions: Drug: AZD4144 Part B
- Part B2 (healthy Japanese participants) placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo Part B

INTERVENTIONS:
Drug: AZD4144 Part A — Part A: Participants will be administered a single oral dose on Day 1.
  Arms: Part A1 (healthy participants) Cohort 1; Part A1 (healthy participants) Cohort 2; Part A1 (healthy participants) Cohort 3; Part A1 (healthy participants) Cohort 4; Part A1 (healthy participants) Cohort 5; Part A1 (healthy participants) Cohort 6; Part A2 (healthy Japanese participants) Cohort 1; Part A2 (healthy Japanese participants) Cohort 2; Part A3 (healthy Chinese participants) Cohort 1
Drug: AZD4144 Part B — Part B: Participants will be administered a single dose on Day 1, and repeated dosing will commence from Day 4 until Day 11 (inclusive) and a single dose on Day 12.
  Arms: Part B1 (healthy participants) Cohort 1; Part B1 (healthy participants) Cohort 2; Part B1 (healthy participants) Cohort 3; Part B2 (healthy Japanese participants) Cohort 1
Drug: Placebo Part A — Part A: Participants will be administered a single oral dose of matching placebo on Day 1.
  Arms: Part A1 (healthy participants) placebo; Part A2 (healthy Japanese participants) placebo; Part A3 (healthy Chinese participants) placebo
Drug: Placebo Part B — Part B: Participants will be administered a single dose of matching placebo on Day 1, and repeated dosing will commence from Day 4 until Day 11 (inclusive) and a single dose on Day 12.
  Arms: Part B1 (healthy participants) placebo; Part B2 (healthy Japanese participants) placebo

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single and multiple ascending doses of AZD4144 administered orally in healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, first time-in human (FTiH), randomised, single-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) sequential group study in healthy participants.

Part A consists of 3 parts:

Part A1 (healthy participants) Part A2 (healthy Japanese participants) and Part A3 (healthy Chinese participants)

Part B consists of 2 parts:

Part B1 (healthy participants) Part B2 (healthy Japanese participants)

Both Part A and Part B of the study will comprise of a screening period of maximum 28 days. The treatment period would last from Day -1 to Day 4 in Part A and from Day -1 to Day 15 in Part B of the study. A follow up visit will be performed on Day 10 + 3 days for Part A and on Day 20 + 3 days for Part B.

Each participant will participate for about 6 weeks in Part A of the study and for about 7 weeks in Part B of the study.

ELIGIBILITY:
Inclusion criteria:

* Females must have a negative pregnancy test, must not be lactating and must be of non-childbearing potential.
* Have a BMI between 18 and 32 kg/m2 inclusive at both Screening and Admission and weigh at least 45 kg at Screening.
* For healthy Japanese cohorts (Part A2 and Part B2): healthy male and female (of non-childbearing potential) participants are to be Japanese, defined as having both parents and four grandparents who are Japanese. This included second and third generation participants of Japanese descent whose parents or grandparents are living in a country other than Japan.
* For healthy Chinese cohort (Part A3): healthy male and female (of non-childbearing potential) Chinese participants for whom both parents and all grandparents are Chinese and not lived outside of China for more than 10 years.

Exclusion criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma.
* Clinically significant serious active and chronic infections.
* Bacillus Calmette-Guérin vaccine within one year prior to signing the ICF.
* Any abnormal laboratory values at the Screening Visit.
* Any positive result on Screening for serum Hepatitis B surface antigen (HBsAg), anti-Hepatitis B core (HBc), hepatitis C antibody, or Human Immunodeficiency Virus (HIV).
* Any cardiac abnormalities.
* History of alcohol abuse or drug abuse.
* Current smokers or those who have smoked or used nicotine products.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Clinical signs and symptoms consistent with COVID-19.
* In addition, any of the following is regarded as a criterion for exclusion from the genetic research:

  1. Previous bone marrow transplant
  2. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Part A: From screening (Day -28 to Day -2) to Day 10; Part B: From screening (Day -28 to Day-2) to Day 20
  To assess the safety and tolerability of AZD4144 following oral administration of single and multiple ascending doses (Part A and Part B)

SECONDARY OUTCOMES:
Maximum observed plasma (peak) drug concentration (Cmax) | Part A: Day 1 to Day 4. and Day 10; Part B: Day 1 to Day 15 and Day 20
  To characterise the single dose and steady state PK of AZD4144 following oral administration of single and multiple ascending doses (Part A and Part B).
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) | Part A: Day 1 to Day 4. and Day 10; Part B: Day 1 to Day 15 and Day 20
  To characterise the single dose and steady state PK of AZD4144 following oral administration of single and multiple ascending doses (Part A and Part B)
Area under plasma concentration-time curve from zero to infinity (AUC0-inf) | Part A: Day 1 to Day 4. and Day 10; Part B: Day 1 to Day 15 and Day 20
  To characterise the single dose and steady state PK of AZD4144 following oral administration of single and multiple ascending doses (Part A and Part B)
Renal clearance of drug from plasma (CLR) | Part A: Day 1 to Day 4. and Day 10; Part B: Day 1 to Day 15 and Day 20
  To characterise the single dose and steady state PK of AZD4144 following oral administration of single and multiple ascending doses (Part A and Part B)
PD analysis: Levels of disease-specific biomarkers | Part A: Day 1 to Day 4 and Day 10; Part B: Day -1, Day 1 to Day 4, Day 12 to Day 15 and Day 20
  To assess the effect of AZD4144 on levels of disease-specific biomarkers.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/